CLINICAL TRIAL: NCT03412045
Title: Hyperbaric Oxygen Therapy in Sickle Cell Pain
Acronym: HAVOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0003-17-FB
Record Dates: First submitted 2017-12-05; First posted 2018-01-26 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-06

CONDITIONS: Vaso-occlusive Crisis; Sickle Cell Anemia Crisis
MeSH Terms: conditions — Vaso-Occlusive Crises | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: This study will use a convenience sample of patients admitted to hospital for vaso-occlusive sickle cell crisis to be treated with hyperbaric oxygen (HBO), the intervention, in an effort to ameliorate pain and shorten the length of hospital stay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- treatment (Experimental): This preliminary study will be a convenience sample of patients admitted to hospital for vaso-occlusive sickle cell crisis to be treated with hyperbaric oxygen (HBO), the intervention, in an effort to ameliorate pain and shorten the length of hospital stay.
  Interventions: Device: hyperbaric oxygen therapy

INTERVENTIONS:
Device: hyperbaric oxygen therapy — Participants in vaso-occlusive crisis from sickle cell anemia will receive 1-3 hyperbaric oxygen (HBO) sessions depending on response to the therapy. Each session will be approximately 2 hours in length at 2.5 ATM. Minimum time between HBO sessions of 4 hours.

SUMMARY:
Sickle cell anemia is a genetic blood disorder where red blood cells are abnormally shaped, crescent- or sickle-shaped, instead of the normal, round shape. This misshapen cell is rigid and sticky, causing them to clump together and block small blood vessels. This blockage can lead to pain, infections, and organ damage, and the shortened lifespan of sickle cells causes anemia. The purpose of this study is to explore if hyperbaric oxygen (HBO) therapy would decrease pain and hospital length of stay associated with acute sickle cell pain crisis. Adults presenting with an uncomplicated acute pain crisis (i.e., acute chest syndrome, acute myocardial infarction/stroke) would be eligible. The intervention would be 1-3 hyperbaric oxygen sessions depending on response to therapy. Each treatment session will be approximately two hours in length. Evaluation would be through participants' self--assessment via the visual analog scale for pain level before and after treatments as well as tracking length of stay in the hospital.

DETAILED DESCRIPTION:
Sickle cell anemia is a genetic blood disorder where red blood cells are abnormally shaped, crescent- or sickle-shaped, instead of the normal, round shape. This misshapen cell is rigid and sticky, causing them to clump together and block small blood vessels. This blockage can lead to pain, infections, and organ damage, and the shortened lifespan of sickle cells causes anemia. Previous study suggest that hyperbaric oxygen (HBO) may help ameliorate symptoms and have positive effects for sickle cell patients. In addition, although a few studies did discuss pain reduction associated with HBO therapy, results are conflicting, and sample sizes are too small to carry any weight when compared against each other. No information has been gathered to date about how HBO therapy this may affect hospital length of stay. The purpose of this study is to determine if HBO treatment in participants experiencing sickle cell crisis would produce a decrease in pain and decrease in hospital length of stay.

Current standard of care at University of Nebraska Medical Center (UNMC) and Nebraska Medicine for patients identified as having sickle cell and experiencing an uncomplicated pain crisis that is not responding to acute treatment in the emergency department over the course of a few hours is to admit the patient to the hematology service. They would receive IV fluid administration, oxygen, and usually large doses of pain medications, until their pain subsides. Patient's complete blood count (CBC) and comprehensive metabolic panel (CMP) are monitored during this time for acute changes. Once pain has subsided and no signs of complications such as infection, etc. are found, the patient is discharged with follow up in hematology clinic.

Interventions would be 1-3 hyperbaric oxygen sessions depending on response to the therapy. Each treatment session will be approximately two hours in length. Evaluation would be through participants' self-assessment via the visual analog scale for pain level before and after treatments as well as tracking length of stay in the hospital. Changes in pain ratings will use the visual pain scale of 0 to 100, where 0 is no pain and 100 being maximal pain imaginable for that participant. Pain ratings will be compiled and compared 1 hour before and after each treatment and from daily pain ratings assessed at hospital admission until discharge. Hospital length of stay is recorded for each participant from date of randomization until date of discharge or date of death from any cause and compared to data extracted from the electronic health record system EPIC.

ELIGIBILITY:
Inclusion Criteria:

* 19 years old or older
* Present with an uncomplicated sickle cell crisis at admission friom the emergency department

Exclusion Criteria:

* < 19 years old
* pregnant female
* complicated sickle cell crisis present (i.e., concomitant MI, stroke, acute chest syndrome at time of presentation)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Pain Assessment per Treatment | one hour before and after each hyperbaric treatment
  Change in pain rating will be determined within one hour before and after each hyperbaric oxygen (HBO) treatment. The pain scale is 0-100, 0 being no pain and 100 being maximal pain imaginable for that participant. Pain assessments before and after each HBO treatment will be compiled and compared to determine treatment effectiveness.

SECONDARY OUTCOMES:
Hospital Length of Stay | up to 1 month
  The hospital length of stay in days from date of randomization until date of discharge or date of death from any cause, whichever came first is recorded and compared to data extracted from the electronic health record system EPIC.
Pain Assessment for All Treatments | up to 1 month (expected average of 3 days)
  Change in pain rating will be determined between enrollment and hospital discharge. The scale is 0-100, 0 being no pain and 100 being maximal pain imaginable for that participant. Pain assessments will occur at initial Emergency Department (ED) presentation and then every morning of admission until discharge. Pain completely resolved or max session number of 3 will be used as standard to halt HBO therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff S Cooper, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT03412045/ICF_001.pdf